CLINICAL TRIAL: NCT05916742
Title: Functionalization of a Volume-stable Collagen Matrix (VCMX) Using Injectable Platelet Rich Fibrin (i-PRF) for the Treatment of Single Gingival Recession
Brief Title: Biofunctionalization of a Volume-stable Collagen Matrix (VCMX) for the Treatment of Single Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Associate professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCMX+iPRF
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Gingival Recession
Keywords: Platelet-rich fibrin; Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Drug Prescriptions; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAF+VCMX+i-PRF (Experimental): The surgical procedure for root coverage will be the trapezoidal-type of coronally advanced flap previously described (de Sanctis & Zucchelli 2007). Thus, it will start with two divergent releasing incisions lateral to the gingival recession defect. These releasing incisions will then be united by a sulcular incision, and the flap will be raised beyond the mucogingival junction. Subsequently, a VCMX functionalized with injectable platelet rich-fibrin (I-PRF) will be placed at the cemento-enamel junction (CEJ) level and stabilized in the adjacent interdental connective beds by interrupted sutures. Then, sling sutures will be placed to stabilize the flap margin 2 mm coronal to CEJ, followed by interrupted sutures to close the releasing incisions.
  Interventions: Procedure: CAF; Procedure: i-PRF; Device: VCMX; Drug: Sodium dipyrone; Drug: Chlorhexidine rinse; Drug: Amoxicillin 500mg
- CAF+VCMX (Experimental): The surgical procedure for root coverage will be the trapezoidal-type of coronally advanced flap previously described (de Sanctis & Zucchelli 2007). Thus, it will start with two divergent releasing incisions lateral to the gingival recession defect. These releasing incisions will then be united by a sulcular incision, and the flap will be raised beyond the mucogingival junction. Subsequently, a VCMX will be placed at the cemento-enamel junction (CEJ) level and stabilized in the adjacent interdental connective beds by interrupted sutures. Then, sling sutures will be placed to stabilize the flap margin 2 mm coronal to CEJ, followed by interrupted sutures to close the releasing incisions.
  Interventions: Procedure: CAF; Device: VCMX; Drug: Sodium dipyrone; Drug: Chlorhexidine rinse; Drug: Amoxicillin 500mg
- CAF (Active Comparator): The surgical procedure for root coverage will be the trapezoidal-type of coronally advanced flap previously described (de Sanctis & Zucchelli 2007). Thus, it will start with two divergent releasing incisions lateral to the gingival recession defect. These releasing incisions will then be united by a sulcular incision, and the flap will be raised beyond the mucogingival junction. Then, sling sutures will be placed to stabilize the flap margin 2 mm coronal to CEJ, followed by interrupted sutures to close the releasing incisions.
  Interventions: Procedure: CAF; Drug: Sodium dipyrone; Drug: Chlorhexidine rinse; Drug: Amoxicillin 500mg

INTERVENTIONS:
Procedure: CAF — Periodontal surgical technique to treat gingival recessions
  Other Names: Periodontal plastic surgery
Procedure: i-PRF — Blood-derived biomaterial. Two sterile plastic tubes (Process for PRF, Nice, France) with a volume of 10 ml will be used to generate fluid blood concentrate. After blood collection, the tubes will be centrifuged using a Duo centrifuge (Process for PRF, Nice, France) (fixed angle rotor with a radius of 110 mm) following the protocol proposed by Choukroun et al. (2018) (600 rpm; 8 min).
  Other Names: injectable platelet rich-fibrin
  Arms: CAF+VCMX+i-PRF
Device: VCMX — Porcine derived collagen matrix.
  Other Names: Volume-stable collagen matrix; Geistlich Fibro-Gide
  Arms: CAF+VCMX; CAF+VCMX+i-PRF
Drug: Sodium dipyrone — All participants will be instructed to take 500 mg sodium dipyrone just in case of pain.
  Other Names: Drug prescription
Drug: Chlorhexidine rinse — All participants will be instructed to perform 0.12% chlorhexidine rinse after the surgical procedures.
  Other Names: Drug prescription
Drug: Amoxicillin 500mg — Participants enrolled in the CAF+VCMX and CAF+VCMX will be instructed to take amoxicillin 500mg (8 hours/8 hours, during 7 days) after the surgical procedures.
  Other Names: Drug prescription

SUMMARY:
The treatment of single gingival recessions comprises different well-established techniques, and the association between coronally advanced flap (CAF) and the subepithelial connective tissue graft is considered the gold standard. However, despite the excellent clinical results obtained, the use of subepithelial connective tissue graft is related to an increased risk of trans and postoperative bleeding, a longer duration of the surgical procedure and greater postoperative pain and morbidity. To overcome these limitations and increase patient acceptance, new biomaterials have been developed as possible alternatives to the use of connective tissue graft. Recently, tissue engineering has been investigating collagen matrices as carriers of biologically active substances. In vitro and in vivo studies have shown that the biofunctionalization of these matrices using injectable platelet rich-fibrin (i-PRF) can optimize the healing process of soft tissues using own's patient regenerative components. However, although it has promising potential, clinical studies evaluating the performance of functionalized collagen matrices are still scarce in the literature. Thus, the present study aims to evaluate the clinical, esthetic, patient-centered, immuno and microbiological results of the use of the biofunctionalized volume stable collagen matrix (VCMX) for the treatment of single gingival recessions RT1. For such purpose, a randomized controlled clinical trial of superiority, parallel and blind will be carried out. Seventy-five patients with RT1 single gingival recession will be selected, who will be randomly allocated to one of the following groups: CAF+VCMX+i-PRF (n = 25), coronally advanced flap associated with VCMX functionalized with i-PRF; CAF+VCMX (n=25), coronally advanced flap associated with VCMX; and CAF group (n = 25), coronally advanced flap alone (CAF). The groups will be compared regarding clinical, esthetic and patient-centered outcomes at the baseline, three and six months after the surgical procedure. The microbiological evaluation will be performed at baseline, three and six months after surgery and the concentration of inflammatory markers and growth factors will be assessed before the procedure and 3, 7, 14, 30 and 60 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of RT1 (Cairo et al., 2011) buccal single gingival recession (GR) on vital upper or lower canines and premolars with intact root surface (visible CEJ).
* Presence of dentin hypersensitivity (HD) and/or esthetic concerns related to GR.
* Adults > 18 years old.
* Systemically health.
* No signs of active periodontal disease.
* Full-mouth plaque and bleeding score ≤ 20%.
* Written informed consent given.

Exclusion Criteria:

* Smoking.
* Contraindication for periodontal surgery.
* Pregnancy.
* Presence of orthodontic braces.
* Medications known to interfere with periodontal healing.
* Use of anticoagulants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-18 (Estimated)

PRIMARY OUTCOMES:
Gingival recession reduction (RecRed) | 6 months
  Final depth of gingival recession in millimeters minus gingival margin initial position in millimeters measured through a periodontal probe.

SECONDARY OUTCOMES:
Root coverage esthetic score | 6 months
  The Root Coverage Esthetic Scale (RES; Cairo et al., 2009) will be performed by two blinded and independent examiners at the 6-month post-operative assessment. This score evaluates five variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color.
Dentine hypersensitivity | 6 months
  Evaluation of root sensitivity with the air blow test and measurement with a visual analog scale (VAS).
Patient recovery | 14 days
  Evaluation of postsurgery sequelae, pain, and discomfort, oral function and interference with daily activities through postoperative diary previously described (Tonetti et al. 2018).
Patient-centred esthetic evaluation | 6 months
  Esthetic evaluation performed by the patient through a visual analog scale (VAS).
Immunological evaluation | Baseline, 3, 7, 14, 30, and 60 days after surgery
  Gingival crevicular fluid will be collected in order to evaluate the levels of nine inflammatory markers: IL1β, IL4, IL5, IL6, IL9, IL10, IL17A, Interferon gamma-induced protein 10 kDa (IP10), macrophage inflammatory protein 1α (MIP1α), monocyte chemotactic protein 1α (MCP-1α), and tumor necrosis factor α (TNFα). The following growth factors will be evaluated: EGF, TGF, PDGF, FGF, and VEGF. In addition, MMP-1, MMP-2 from TIMP-1, and TIMP-2 will also be evaluated.
Microbiological evaluation | Baseline, 45 days, and 6 months after the procedure.
  The collection of the subgingival biofilm will be performed in order to quantificate microorganisms such as Porphyromonas gingivalis, Tannerella forsythia, Prevotella intermedia, Fusobacterium nucleatum e Streptococcus sanguinis.

CONTACTS AND LOCATIONS:
Locations (1):
- São Paulo State University, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tonetti MS, Cortellini P, Pellegrini G, Nieri M, Bonaccini D, Allegri M, Bouchard P, Cairo F, Conforti G, Fourmousis I, Graziani F, Guerrero A, Halben J, Malet J, Rasperini G, Topoll H, Wachtel H, Wallkamm B, Zabalegui I, Zuhr O. Xenogenic collagen matrix or autologous connective tissue graft as adjunct to coronally advanced flaps for coverage of multiple adjacent gingival recession: Randomized trial assessing non-inferiority in root coverage and superiority in oral health-related quality of life. J Clin Periodontol. 2018 Jan;45(1):78-88. doi: 10.1111/jcpe.12834. Epub 2017 Nov 21. PMID 29087001
- [Background] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093
- [Background] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597
- [Background] Choukroun J, Ghanaati S. Reduction of relative centrifugation force within injectable platelet-rich-fibrin (PRF) concentrates advances patients' own inflammatory cells, platelets and growth factors: the first introduction to the low speed centrifugation concept. Eur J Trauma Emerg Surg. 2018 Feb;44(1):87-95. doi: 10.1007/s00068-017-0767-9. Epub 2017 Mar 10. PMID 28283682